CLINICAL TRIAL: NCT04831645
Title: The Use of a Dynamic Sustained Compression Intramedullary Nail for Tibiotalocalcaneal Arthrodesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MedShape, Inc (Industry)
Collaborators: CurveBeam LLC (Unknown); Orthopedic Foot and Ankle Center, Ohio (Other)
Responsible Party: Sponsor
Other Study IDs: MedShape011221
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-04

CONDITIONS: Ankle Arthritis; Arthritis Foot
Keywords: Subtalar Arthrodesis; Intramedullary Nail; Ankle Arthrodesis; Internal Fixation; Sustained Compression; Longitudinal Computed Tomography; Tibiotalar Arthrodesis; Joint Fusion
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: DynaNail — Utilization of a novel dynamic compression pseudoelastic intramedullary nail
Procedure: Tibiotalocalcaneal Arthrodesis — Tibiotalocalcaneal (TTC) arthrodesis with a novel dynamic compression intramedullary nail.
  Other Names: Subtalar Arthrodesis; Tibiotalar Arthrodesis

SUMMARY:
The purpose of this study is to determine the clinical efficacy of a novel sustained dynamic compression intramedullary nail for tibiotalocalcaneal (TTC) arthrodesis utilizing longitudinal weight-bearing computed tomographic imaging. Of particular focus will be assessment of compressive element recovery and its relation to fusion development over time and weight-bearing status. Additionally, the study will incorporate longitudinal fusion assessment to evaluate differences between three-dimensional weight-bearing computed tomography (WBCT) scans and two-dimensional radiographs (X-rays) at multiple points of the fusion process. Finally, the study will evaluate the differences in WBCT-based fusion assessment between automated and manual methodologies for fusion area calculation.

DETAILED DESCRIPTION:
This study is a collaborative effort between the Orthopedic Foot and Ankle Center, MedShape, Inc, and CurveBeam. This is a prospective investigation to assess the clinical outcomes of patients with a tibiotalocalcaneal arthrodesis with the Sustained Dynamic Compression Intramedullary Nail (DynaNail), including longitudinal assessment with weight-bearing CT. The investigators plan to enroll 45 patients. No placebo control will be used, as there is no other IM nail available capable of providing sustained compression. Additionally, given that many patients receiving this treatment have had prior failed treatments and face poor alternatives such as amputation, using a prior-generation IM nail as a control treatment would be unethical.

Design:

This is a prospective, single-group study. Patients of the Orthopedic Foot and Ankle Center who are scheduled to undergo TTC arthrodesis will be screened for eligibility and informed consent will be obtained from those who meet the inclusion/exclusion criteria. Subjects will be assessed pre-operatively and then at five post-operative intervals: 1 week, 6 weeks, 3 months, 6 months, and 12 months. A WBCT scan will be obtained at each interval.

Selection of Subjects:

Patients will be identified in the clinic by an attending orthopaedic foot and ankle surgeon or his/her physician assistant based on clinical exam and radiographic findings. Patients will be screened for eligibility by the research coordinator/ key personnel in close coordination with the surgeon and co-investigator.

Pre-operative Questionnaire:

After informed consent, the patients will be asked to complete patient reported outcomes questionnaires that are part of the SOS Registry associated with function and pain, including VAS, VR-12, FFI-R, FAAM, AOS, and AOFAS. The patients will also be asked to provide information related to prior medical history (including potential co-morbidities associated with non-union, i.e. tobacco usage, neuropathy, renal disease, obesity, etc.) and surgical history of the subject lower extremity.

Surgery:

The following surgical procedure is standard of care. The surgical procedure will involve both tibiotalar and talocalcaneal joint preparation through any approach (lateral, posterior, anterior with sinus tarsi). The use of supplemental bone graft is at the discretion of the treating surgeon but must be documented. The MedShape DynaNail will then be inserted according to the manufacturer's technique. The patient will be placed in a short leg splint and kept non-weight bearing initially. The patient will be discharged from the hospital when medically ready. Weight-bearing will start at seven weeks post-surgery.

Follow-Up Visits and Questionnaires:

The patient will return to clinic for visits at the following intervals after surgery: 1 week, 6 weeks, 3 months, 6 months, and 12 months. At each of these time points, a clinical exam will be conducted, and SOS patient questionnaires will be administered, as well as a radiographic and clinical follow-up form. Additionally, radiograph and weight-bearing CT imaging will be obtained of both the ankle and subtalar joints. At 3 months and 12 months post-op, all X-ray and CT images will be de-identified, burned to a DVD, and copies will be sent to both co-sponsors.

ELIGIBILITY:
Inclusion Criteria:

* Meets indications for TTC arthrodesis and receives the DynaNail implant
* Able to understand the requirements of the study
* Willing to comply with the study protocol
* Sign an Informed consent
* 18 years of age or older

Exclusion Criteria:

* Investigator determines that the subject is unlikely to comply with the requirements of the study
* Non-English speaker
* Blind
* Illiterate
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Orthopedic Foot and Ankle Center with end-stage tibiotalar (ankle) and talocalcaneal (subtalar) joint arthritis from any etiology will be eligible to enroll in the study. In general, tibiotalar and subtalar arthritis is caused by trauma. Traumatic injuries have no predilection for race, religion, cultural background, etc. Therefore, all demographic groups will have access to this study and should be represented.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2024-05-24 (Estimated); Study Completion 2024-05-24 (Estimated)

PRIMARY OUTCOMES:
Fusion | Pre-Operative to 1 year post-surgery
  Joint Fusion, as measured by radiographs and CT scans. Fusion rates will be assessed based on varying CT fusion areas. Fusion rates based on X-Ray vs CT assessment will also be compared. CT fusion rates based on varying fusion areas will be compared with PROM data to assess which fusion area actually corresponds to increased function and reduced pain.

SECONDARY OUTCOMES:
VAS | Pre-Operative up to one year post-surgery
  Visual Analog Scaled (VAS) - Rates the intensity of pain from 0 - 10 with 10 being the worst pain possible and 0 being no pain.
VR-12 | Pre-Operative up to one year post-surgery
  The Veterans RAND 12 Item Health Survey (VR-12, formerly called the Veterans SF-12) was developed from the Veterans RAND 36 (VR-36, formerly called the Veterans SF-36), which was modified from the original MOS SF-36. The VR-12 measures Physical functioning (PF), social functioning (SF), role limitation due to physical problems (RP), role limitation due to emotional problems (RE), mental health (MH), energy and vitality (VT), bodily pain (BP) and general perception of health (GH). Standard based scoring (sometimes called norm based scoring) is used to calculate the physical component summary (PCS) and mental component summary (MCS) for both measures. The PCS and MCS are standardized using a t-score transformation and normed to a US population at a score of 50 and a standard deviation of 10. Higher scores indicate better health.
FFI-R | Pre-Operative up to one year post-surgery
  Foot Function Index-Revised - Measures the impact of foot pathology on function in terms of pain, disability, and activity restriction. The score is a percentage. The higher the score, the greater the disability.
FAAM | Pre-Operative up to one year post-surgery
  Foot and Ankle Ability Measure - Measures patient capacity for sports and activities of daily living (ADL). The final score is a percentage. The higher final score represents a higher level of physical function.
AOS | Pre-Operative up to one year post-surgery
  Ankle Osteoarthritis Scale - Measures pain levels and difficulty performing various activities of daily living. A line-based scale with range from no pain to the worst pain imaginable.
AOFAS | Pre-Operative up to one year post-surgery
  American Orthopaedic Foot and Ankle Society Scale - Clinician-based outcome that measures foot/ankle pain, function, and alignment. The lower the score, the greater the disability. The maximum score is 100.

OTHER OUTCOMES:
Automated vs Manual Fusion Assessment | Up to one year post-surgery
  Fusion area calculation over time will be assessed not only by two clinically-trained reviewers, but also using CurveBeam's automated CubeVue assessment software. Averaged clinician results will be compared with CubeVue-calculated data.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Berlet, MD, Principal Investigator — Orthopedic Foot and Ankle Center
Locations (1):
- Orthopedic Foot and Ankle Center, Worthington, Ohio, United States

IPD SHARING:
Plan to Share IPD: No